CLINICAL TRIAL: NCT02350673
Title: A Phase 1b, Open-Label, Multi-Center, Dose Escalation Study of the Safety, Pharmacokinetics, and Therapeutic Activity of Cergutuzumab Amunaleukin, an Immunocytokine, Which Consists of a Variant of Interleukin 2 (IL 2v), That Targets Carcinoembryonic Antigen (CEA), and Atezolizumab, an Antibody That Targets Programmed Death-Ligand 1 (PD-L1), Administered Intravenously, in Patients With Locally Advanced and/or Metastatic Solid Tumors
Brief Title: A Study of Intravenous (IV) Cergutuzumab Amunaleukin and Atezolizumab in Combination in Participants With Locally Advanced and/or Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BP29435; 2014-000948-14 (EudraCT Number)
Record Dates: First submitted 2015-01-20; First posted 2015-01-30 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Solid Tumors
MeSH Terms: interventions — atezolizumab

ARMS (2):
- Cergutuzumab+Atezolizumab (Part I) (Experimental): Participants will receive escalated IV doses of cergutuzumab amunaleukin in combination with atezolizumab. This is a Part I dose escalation phase of the study. Cergutuzumab amunaleukin will be escalated from a starting dose of 6 milligrams (mg) and dosing schedules of every week (qw) and every 2 weeks (q2w) may be explored. Atezolizumab will be administered in fixed flat doses of either 840 mg q2w or 1200 mg every 3 weeks (q3w). Treatment will be continued until loss of clinical benefit, unacceptable toxicities, or withdrawal of consent for a maximum treatment period of 24 months for both cergutuzumab amunaleukin and atezolizumab and may be modified if emerging data suggest longer treatment period is needed.
  Interventions: Drug: Atezolizumab; Drug: Cergutuzumab Amunaleukin
- Cergutuzumab +Atezolizumab (Part II) (Experimental): This is a Part II expansion phase of the study. Participants will receive cergutuzumab amunaleukin at maximum tolerated dose (MTD) (or recommended dose) identified during Part I in combination with atezolizumab. Treatment will be continued until loss of clinical benefit, unacceptable toxicities, or withdrawal of consent for a maximum treatment period of 24 months for both cergutuzumab amunaleukin and atezolizumab and may be modified if emerging data suggest longer treatment period is needed.
  Interventions: Drug: Atezolizumab; Drug: Cergutuzumab Amunaleukin

INTERVENTIONS:
Drug: Atezolizumab — Participants will receive atezolizumab IV infusion at doses of 800 mg q2w or 1200 mg q3w.
  Other Names: MPDL3280A, Tecentriq®
Drug: Cergutuzumab Amunaleukin — Participants will receive cergutuzumab amunaleukin IV infusion at escalated doses and at different dosing schedules in Part I and at MTD (or recommended dose) in Part II.
  Other Names: RO6895882, CEA-IL2v

SUMMARY:
This is an open-label, multi-center, Phase Ib clinical study of cergutuzumab amunaleukin, in combination with atezolizumab, to investigate the safety, pharmacokinetics, and therapeutic activity in participants with locally advanced and/or metastatic carcinoembryonic antigen (CEA)-positive solid tumors, whose disease has progressed on or who are intolerant to the standard of care therapy. Enrolled participants who continue treatment will be treated until loss of clinical benefit, unacceptable toxicities, or withdrawal of consent. The study will include 2 parts: a dose-escalation Part I and a dose expansion Part II. The anticipated treatment period is 24 months for both cergutuzumab amunaleukin and atezolizumab and may be modified if emerging data suggest a benefit.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed locally advanced and/or metastatic solid tumor, with at least one tumor lesion of non-critical location accessible to biopsy (with exception of non-small cell lung cancer [NSCLC] participants), and with confirmed progression at baseline that has progressed on, or participant is intolerant to, the standard of care therapy
* Radiologically measurable and clinically evaluable disease as per RECIST v1.1
* Life expectancy, in the opinion of the investigator, greater than or equal to (>=) 12 weeks
* Eastern Cooperative Oncology Group Performance Status 0-1
* All acute toxic effects of any prior radiotherapy, chemotherapy, or surgical procedure must have resolved to Grade less than or equal to (<=) 1, except alopecia (any grade) and Grade 2 peripheral neuropathy
* Adequate cardiac, hematological, liver and renal function
* Negative serum pregnancy test within 7 days prior to study treatment in premenopausal women and women <= 2 years after menopause
* For women who are not postmenopausal and have not undergone surgical sterilization: agreement to remain abstinent or use two adequate non-hormonal methods of contraception including at least one method with a failure rate of <1% per year during the treatment period and for at least five months after the last dose of atezolizumab and at least four months after the last dose of cergutuzumab amunaleukin, whichever is the longest
* For men: agreement to remain abstinent or use contraceptive measures and agreement to refrain from donating sperm
* Locally or centrally confirmed CEA expression in archival tumor tissue
* Participants with unilateral pleural effusion will be eligible for inclusion if they fulfill the Global Initiative for Obstructive Lung Disease classification of 0-1 level for pulmonary function and New York Heart Association (NYHA) classification class 1 for cardiac function

Exclusion Criteria:

* Active or untreated central nervous system (CNS) metastases as determined by computed tomography (CT) or magnetic resonance imaging evaluation during screening and prior radiographic assessments; participants with a history of treated asymptomatic CNS metastases are eligible
* Spinal cord compression not definitively treated with surgery and/or radiation or previously diagnosed and treated spinal cord compression without evidence that disease has been clinically stable for >= 2 weeks prior to randomization
* Leptomeningeal disease
* Participants with an active second malignancy (other than non-melanoma skin cancer or cervical carcinoma in situ). Participants who have a history of malignancy are not considered to have an active malignancy if they have completed therapy and are considered by their treating physician to be at <= 30 percent (%) risk for relapse
* Evidence of significant, uncontrolled concomitant diseases which could affect compliance with the protocol or interpretation of results, including diabetes mellitus, history of relevant pulmonary disorders, and known autoimmune diseases
* Participants with bilateral pleural effusion and NSCLC participants with uni- or bilateral effusion confirmed at screening by X-ray are not eligible
* Uncontrolled hypertension, unstable angina, congestive heart failure of any NYHA classification stage greater than (>) 2, serious cardiac arrhythmia requiring treatment (exceptions: atrial fibrillation, paroxysmal supraventricular tachycardia), history of myocardial infarction within 6 months of enrollment
* Administration of a live, attenuated vaccine within 4 weeks before Cycle 1, Day 1 or anticipation that such a live attenuated vaccine will be required during the study. Influenza vaccination should be given during influenza season only. Participants must not receive live, attenuated influenza vaccine within 4 weeks prior to Cycle 1, Day 1, at any time during the study or 5 months after the last dose of atezolizumab
* Known Human Immunodeficiency Virus (HIV)
* Active hepatitis B (HBV) or hepatitis C (HCV) infection
* Severe infections within 4 weeks prior to Cycle 1, Day 1, including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia
* Received oral or intravenous (IV) antibiotics within 2 weeks prior to Cycle 1, Day 1. Participants receiving prophylactic antibiotics (for prevention of a urinary tract infection chronic obstructive pulmonary disease) are eligible
* Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that would contraindicate the use of an investigational drug
* Major surgery or significant traumatic injury less than (<) 28 days prior to the first cergutuzumab amunaleukin infusion (excluding biopsies) or anticipation of the need for major surgery during study treatment
* Dementia or altered mental status that would prohibit informed consent
* History or risk of autoimmune disease, including but not limited to systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Bell's palsy, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis
* Participants with a history of autoimmune hypothyroidism on a stable dose of thyroid replacement hormone or participants with controlled Type 1 diabetes mellitus on a stable insulin regimen may be eligible for this study with approval by the medical monitor
* Inclusion of participants with confirmed positive serology of at least one auto-antibody panel (anti-nuclear antibody, anti-double stranded DNA, cytoplasmic anti-neutrophil cytoplasmic antibody, and perinuclear anti-neutrophil cytoplasmic antibody) at screening should be discussed between Sponsor and investigators, and if judged clinically relevant could be referred to a specialist (Rheumatologist) to exclude an underlying auto-immune disease
* History of idiopathic pulmonary fibrosis, pneumonitis (including drug induced), organizing pneumonia (bronchiolitis obliterans, cryptogenic organizing pneumonia), or evidence of active pneumonitis on screening chest CT scan. History of radiation pneumonitis in the radiation field (fibrosis) is permitted
* Baseline QTc interval > 470 milliseconds (ms), baseline resting bradycardia <45 beats per minute (bpm), or baseline resting tachycardia >100 bpm
* Pregnant or breast-feeding women
* Known hypersensitivity to any of the components of cergutuzumab amunaleukin and atezolizumab; hypersensitivity to Chinese hamster ovary cell products or other recombinant human antibodies
* Investigational therapy within 28 days prior to initiation of study treatment
* Any approved anti-cancer therapy, including chemotherapy or hormonal therapy, within 3 weeks prior to initiation of study treatment, with the exceptions stated in the protocol
* Prior corticosteroids as anti-cancer therapy within a minimum of 14 days of first receipt of study drug
* Last dose with any of the following agents including but not limited to: etanercept, infliximab, tacrolimus, cyclosporine, mycophenolic acid, alefacept, or efalizumab <28 days prior to first dose of study drug
* Last dose of prior immunotherapies including but not limited to: interferon alpha, interferon-beta, interleukin (IL)-2, conjugated IL-2, cergutuzumab amunaleukin (CEA-IL2v) , cytokines, anti-cytotoxic T lymphocyte antigen-4, anti-PD-L1, or anti-PD-1 <28 days prior to first cergutuzumab amunaleukin infusion
* History of severe immune-related adverse effects from CEA-IL2v or anti-PD-1 (nivolumab, pembrolizumab) or anti-PD-L1 (atezolizumab) therapies (Common Terminology Criteria for Adverse Events Grade 3 and 4)
* Regular immunosuppressive therapy
* Treatment with systemic immunosuppressive medications including, but not limited to: prednisone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor agents within 2 weeks prior to Cycle 1, Day 1. Participants who have received acute and/or low-dose systemic immunosuppressant medications may be enrolled in the study after discussion with and approval by the Medical Monitor. The use of inhaled corticosteroids and mineralocorticoids for participants with orthostatic hypotension or adrenocortical insufficiency is allowed
* Radiotherapy within the last 4 weeks before start of study drug treatment with the exception of limited field palliative radiotherapy for bone pain relief

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2015-06-29 (Actual); Primary Completion 2019-12-16 (Actual); Study Completion 2019-12-16 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Dose-Limiting Toxicities | Day 1 up to Day 21
MTD of Cergutuzumab Amunaleukin | Day 1 up to Day 21
Recommended Phase II Dose of Cergutuzumab Amunaleukin | Day 1 up to Day 21
Percentage of Participants with Adverse Events | Baseline up to 30 months
Percentage of Participants with Infusion-Related Reactions | Baseline up to 30 months
Percentage of Participants with Seroconversion of Autoantibodies | Screening up to 30 months (assessed at Screening, predose [Hour 0] on Day 1 of Cycles 2, 4, and 6, and every 3 months after Cycle 6 up to approximately 30 months [cycle length= 14 or 21 days])
  Seroconversion is defined as the presence of at least one of the following autoantibodies: anti-nuclear antibody, antidouble-stranded deoxyribose nucleic acid (DNA), cytoplasmic anti-neutrophil cytoplasmic antibody, and perinuclear anti-neutrophil cytoplasmic antibody.
Forced Expiratory Volume | Screening (up to 28 days prior to Cycle 1 Day 1)
Forced Vital Capacity | Screening (up to 28 days prior to Cycle 1 Day 1)
Percentage of Participants with Anti-Atezolizumab Antibodies | Day 1 Cycle 1 up to 30 months (assessed at Day 1 of Cycles 1, 2, 3, 4, study completion/early discontinuation [up to 30 months], 28 and 120 days post last infusion up to approximately 30 months [cycle length = 14 or 21 days])
Percentage of Participants with Anti-Cergutuzumab Amunaleukin Antibodies | Day 1 Cycle 1 up to 30 months (assessed at Day 1 of Cycles 1, 2, 3, 4, study completion/early discontinuation [up to 30 months], 28 and 120 days post last infusion up to approximately 30 months [cycle length = 14 or 21 days])

SECONDARY OUTCOMES:
Percentage of Participants with Objective Response of Complete Response (CR) or Partial Response (PR) Based on Response Evaluation Criteria in Solid Tumors (RECIST) Version (v) 1.1 as Determined by the Investigator | Screening up to disease progression or death due to any cause whichever occurs first (assessed at Weeks 8 and 12, every 8 weeks thereafter for the first year, and every 12 weeks thereafter up to approximately 30 months overall)
Percentage of Participants with Disease Control (Tumor Response of CR or PR or Stable Disease [SD]) Based on RECIST v1.1 as Determined by the Investigator | Screening up to disease progression or death due to any cause whichever occurs first (assessed at Weeks 8 and 12, every 8 weeks thereafter for the first year, and every 12 weeks thereafter up to approximately 30 months overall)
Percentage of Participants with SD, Based on RECIST v1.1 as Determined by the Investigator | Screening up to disease progression or death due to any cause whichever occurs first (assessed at Weeks 8 and 12, every 8 weeks thereafter for the first year, and every 12 weeks thereafter up to approximately 30 months overall)
Progression-Free Survival Based on RECIST v1.1 as Determined by the Investigator | Screening up to disease progression or death due to any cause whichever occurs first (assessed at Weeks 8 and 12, every 8 weeks thereafter for the first year, and every 12 weeks thereafter up to approximately 30 months overall)
Overall Survival | Screening up to death due to any cause (up to approximately 30 months overall)
Area Under the Concentration Time Curve (AUC) of Cergutuzumab Amunaleukin in "Atezolizumab q2w and Cergutuzumab Amunaleukin q2w" | Baseline up to 30 months (detailed timeframe is provided in the outcome description)
  Atezolizumab is presented as PDL and cergutuzumab amunaleukin as CergA. Pre-infusion (PrI) (Hour 0) of PDL (PDL infusion length=60 minutes [min]), mid of infusion of CergA (CergA infusion length=360 min), end of infusion (EoI), 2, 4, 24, 72, 120 hr after CergA EoI, 169.5 hr after PDL EoI on Day 1, Cycles 1 and 4; 2, 24 hr after CergA EoI on Day 1, Cycle 2; 2 hr after CergA EoI on Day 1, Cycle 3; mid of infusion of CergA, CergA EoI, and 2 hr after CergA EoI infusion on Day 1, Cycle 5; 2, 24, 120 hr after CergA EoI on Day 1, Cycle 6; mid of infusion of CergA, CergA EoI, 2 hr after EoI of CergA on Cycle 7 Day 1 and every cycle thereafter up to study completion/early termination (up to 30 months); 28, 120 days after last infusion (up to 30 months) (cycle length = 14 days)
AUC of Cergutuzumab Amunaleukin in "Atezolizumab q3w and Cergutuzumab Amunaleukin qw" | Baseline up to 30 months (detailed timeframe is provided in the outcome description)
  Atezolizumab is presented as PDL and cergutuzumab amunaleukin as CergA. PrI (Hour 0) of CergA (infusion length=360 min), mid of infusion of CergA, EoI, 1.5, 4, 24, 48, 72, 96 hr after CergA EoI on Day 1, Cycles 1, 2; mid of infusion of CergA, EoI, 1.5, 2, 4, 24, 48, 72, 96 hr after CergA EoI on Days 8 and 15, Cycle 1; 2, 24 hr after CergA EoI on Day 8, Cycle 2; 2 hr after CergA EoI on Day 1, Cycle 3; mid of infusion of CergA, EoI, 2 hr after CergA EoI on Day 15, Cycle 3; 2 hr after CergA EoI on Days 1, 8 Cycle 4; mid of infusion of CergA, EoI, 2 hr after EoI of CergA on Cycle 5 Day 1 and every cycle thereafter up to study completion/early discontinuation (up to 30 months); 28, 120 days after last infusion (up to 30 months) (cycle length = 21 days)
Minimum Drug Concentration (Cmin) of Cergutuzumab Amunaleukin in "Atezolizumab q2w and Cergutuzumab Amunaleukin q2w" | Baseline up to 30 months (detailed timeframe is provided in the outcome description)
  Atezolizumab is presented as PDL and cergutuzumab amunaleukin as CergA. PrI (Hour 0) of PDL (PDL infusion length=60 min), mid of infusion of CergA (CergA infusion length=360 min), EoI, 2, 4, 24, 72, 120 hr after CergA EoI, 169.5 hr after PDL EoI on Day 1, Cycles 1 and 4; 2, 24 hr after CergA EoI on Day 1, Cycle 2; 2 hr after CergA EoI on Day 1, Cycle 3; mid of infusion of CergA, CergA EoI, and 2 hr after CergA EoI infusion on Day 1, Cycle 5; 2, 24, 120 hr after CergA EoI on Day 1, Cycle 6; mid of infusion of CergA, CergA EoI, 2 hr after EoI of CergA on Cycle 7 Day 1 and every cycle thereafter up to study completion/early termination (up to 30 months); 28, 120 days after last infusion (up to 30 months) (cycle length = 14 days)
Cmin of Cergutuzumab Amunaleukin in "Atezolizumab q3w and Cergutuzumab Amunaleukin qw" | Baseline up to 30 months (detailed timeframe is provided in the outcome description)
  Atezolizumab is presented as PDL and cergutuzumab amunaleukin as CergA. PrI (Hour 0) of CergA (infusion length=360 min), mid of infusion of CergA, EoI, 1.5, 4, 24, 48, 72, 96 hr after CergA EoI on Day 1, Cycles 1, 2; mid of infusion of CergA, EoI, 1.5, 2, 4, 24, 48, 72, 96 hr after CergA EoI on Days 8 and 15, Cycle 1; 2, 24 hr after CergA EoI on Day 8, Cycle 2; 2 hr after CergA EoI on Day 1, Cycle 3; mid of infusion of CergA, EoI, 2 hr after CergA EoI on Day 15, Cycle 3; 2 hr after CergA EoI on Days 1, 8 Cycle 4; mid of infusion of CergA, EoI, 2 hr after EoI of CergA on Cycle 5 Day 1 and every cycle thereafter up to study completion/early discontinuation (up to 30 months); 28, 120 days after last infusion (up to 30 months) (cycle length = 21 days)
Maximum Drug Concentration (Cmax) of Cergutuzumab Amunaleukin in "Atezolizumab q2w and Cergutuzumab Amunaleukin q2w" | Baseline up to 30 months (detailed timeframe is provided in the outcome description)
  Atezolizumab is presented as PDL and cergutuzumab amunaleukin as CergA. PrI (Hour 0) of PDL (PDL infusion length=60 min), mid of infusion of CergA (CergA infusion length=360 min), EoI, 2, 4, 24, 72, 120 hr after CergA EoI, 169.5 hr after PDL EoI on Day 1, Cycles 1 and 4; 2, 24 hr after CergA EoI on Day 1, Cycle 2; 2 hr after CergA EoI on Day 1, Cycle 3; mid of infusion of CergA, CergA EoI, and 2 hr after CergA EoI infusion on Day 1, Cycle 5; 2, 24, 120 hr after CergA EoI on Day 1, Cycle 6; mid of infusion of CergA, CergA EoI, 2 hr after EoI of CergA on Cycle 7 Day 1 and every cycle thereafter up to study completion/early termination (up to 30 months); 28, 120 days after last infusion (up to 30 months) (cycle length = 14 days)
Cmax of Cergutuzumab Amunaleukin in "Atezolizumab q3w and Cergutuzumab Amunaleukin qw" | Baseline up to 30 months (detailed timeframe is provided in the outcome description)
  Atezolizumab is presented as PDL and cergutuzumab amunaleukin as CergA. PrI (Hour 0) of CergA (infusion length=360 min), mid of infusion of CergA, EoI, 1.5, 4, 24, 48, 72, 96 hr after CergA EoI on Day 1, Cycles 1, 2; mid of infusion of CergA, EoI, 1.5, 2, 4, 24, 48, 72, 96 hr after CergA EoI on Days 8 and 15, Cycle 1; 2, 24 hr after CergA EoI on Day 8, Cycle 2; 2 hr after CergA EoI on Day 1, Cycle 3; mid of infusion of CergA, EoI, 2 hr after CergA EoI on Day 15, Cycle 3; 2 hr after CergA EoI on Days 1, 8 Cycle 4; mid of infusion of CergA, EoI, 2 hr after EoI of CergA on Cycle 5 Day 1 and every cycle thereafter up to study completion/early discontinuation (up to 30 months); 28, 120 days after last infusion (up to 30 months) (cycle length = 21 days)
Cmin of Atezolizumab in "Atezolizumab q2w and Cergutuzumab Amunaleukin q2w" | Baseline up to 30 months (detailed timeframe is provided in the outcome description)
  Atezolizumab is presented as PDL and cergutuzumab amunaleukin as CergA. PrI (Hour 0) of PDL (PDL infusion length=60 min), mid of infusion of PDL, 0.5, 25.5, 121.5, 169.5, 313.5 hr after EoI of PDL on Day 1, Cycle 1; PrI (Hour 0), mid of infusion, 0.5 and 169.5 hr after PDL EoI on Day 1, Cycle 2; PrI (Hour 0) of PDL on Day 1, Cycle 3; PrI (Hour 0) of PDL, mid of infusion, 0.5, 25.5, 121.5, 169.5, 313.5 hr after PDL EoI on Day 1, Cycles 4, 6; study completion/early termination (up to 30 months), 28 and 120 days after last infusion (up to 30 months) (cycle length = 14 days)
Cmin of Atezolizumab in"Atezolizumab q3w and Cergutuzumab Amunaleukin qw" | Baseline up to 30 months (detailed timeframe is provided in the outcome description)
  Atezolizumab is presented as PDL and cergutuzumab amunaleukin as CergA. PrI (Hour 0) of PDL (PDL infusion length=60 min), mid of infusion of PDL, 0.5, 25.5, 121.5, 169.5 hr after PDL EoI on Day 1, Cycle 1, PrI (Hour 0) of CergA, 72 hr after CergA EoI on Day 15, Cycle 1; PrI (Hour 0) of PDL, mid of infusion of PDL, 0.5, 25.5, 169.5 hr after PDL EoI on Day 1, Cycle 2; 24 hr after CergA administration on Day 9, Cycle 2; PrI (Hour 0) of CergA on Day 15, Cycle 2; PrI (Hour 0) of PDL, 72 hr after CergA EoI, 169.5 hr after PDL EoI on Day 1, Cycle 3, PrI (Hour 0) of PDL on Day 15, Cycle 3; PrI (Hour 0) of PDL, mid of infusion of PDL, 0.5, 169.5 hr after PDL EoI on Day 1, Cycle 4; study completion/early termination (up to 30 months), 28 and 120 days after last infusion (up to 30 months) (cycle length = 21 days)
Cmax of Atezolizumab in "Atezolizumab q2w and Cergutuzumab Amunaleukin q2w" | Baseline up to 30 months (detailed timeframe is provided in the outcome description)
  Atezolizumab is presented as PDL and cergutuzumab amunaleukin as CergA. PrI (Hour 0) of PDL (PDL infusion length=60 min), mid of infusion of PDL, 0.5, 25.5, 121.5, 169.5, 313.5 hr after EoI of PDL on Day 1, Cycle 1; PrI (Hour 0), mid of infusion, 0.5 and 169.5 hr after PDL EoI on Day 1, Cycle 2; PrI (Hour 0) of PDL on Day 1, Cycle 3; PrI (Hour 0) of PDL, mid of infusion, 0.5, 25.5, 121.5, 169.5, 313.5 hr after PDL EoI on Day 1, Cycles 4, 6; study completion/early termination (up to 30 months), 28 and 120 days after last infusion (up to 30 months) (cycle length = 14 days)
Cmax of Atezolizumab in "Atezolizumab q3w and Cergutuzumab Amunaleukin qw" | Baseline up to 30 months (detailed timeframe is provided in the outcome description)
  Atezolizumab is presented as PDL and cergutuzumab amunaleukin as CergA. PrI (Hour 0) of PDL (PDL infusion length=60 min), mid of infusion of PDL, 0.5, 25.5, 121.5, 169.5 hr after PDL EoI on Day 1, Cycle 1, PrI (Hour 0) of CergA, 72 hr after CergA EoI on Day 15, Cycle 1; PrI (Hour 0) of PDL, mid of infusion of PDL, 0.5, 25.5, 169.5 hr after PDL EoI on Day 1, Cycle 2; 24 hr after CergA administration on Day 9, Cycle 2; PrI (Hour 0) of CergA on Day 15, Cycle 2; PrI (Hour 0) of PDL, 72 hr after CergA EoI, 169.5 hr after PDL EoI on Day 1, Cycle 3, PrI (Hour 0) of PDL on Day 15, Cycle 3; PrI (Hour 0) of PDL, mid of infusion of PDL, 0.5, 169.5 hr after PDL EoI on Day 1, Cycle 4; study completion/early termination (up to 30 months), 28 and 120 days after last infusion (up to 30 months) (cycle length = 21 days)
Change from Baseline in Cluster of Differentiation (CD) 4 Positive (+) Type of Lymphocytes | From Baseline to 30 months
Change from Baseline in CD8+ Type of Lymphocytes | From Baseline to 30 months
Change from Baseline in Natural Killer Cells | From Baseline to 30 months
Change from Baseline in Monocytes | From Baseline to 30 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (14):
- United States (4):
  - Yale Cancer Center; Medical Oncology, New Haven, Connecticut
  - Columbia Univ Med Ctr, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - SCRI-Tennessee Oncology, Nashville, Tennessee
- University Health Network; Princess Margaret Hospital; Medical Oncology Dept, Toronto, Ontario, Canada
- Denmark (2):
  - Herlev Hospital; Onkologisk afdeling, Herlev
  - Rigshospitalet; Onkologisk Klinik, København Ø
- Netherlands (2):
  - Antoni van Leeuwenhoek Ziekenhuis, Amsterdam
  - Erasmus MC, Rotterdam
- Spain (4):
  - Clinica Universitaria de Navarra; Servicio de oncología, Pamplona, Navarre
  - Hospital Univ Vall d'Hebron; Servicio de Oncologia, Barcelona
  - START Madrid. Centro Integral Oncologico Clara Campal; CIOCC, Madrid
  - Hospital Clinico Universitario de Valencia; Servicio de Onco-hematologia, Valencia
- CHUV; Departement d'Oncologie, Lausanne, Switzerland